CLINICAL TRIAL: NCT01781611
Title: Dipyridamole Assessment for Flare Reduction in SLE
Brief Title: Dipyridamole Assessment for Flare Reduction in Systemic Lupus Erythematosus (SLE)
Acronym: DARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Oklahoma Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB# 12-10
Record Dates: First submitted 2013-01-02; First posted 2013-02-01 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus; dipyridamole
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Aspirin; Aspirin, Dipyridamole Drug Combination

STUDY DESIGN:
Intervention Model Description: Pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- extended release dipyridamole/aspirin (Experimental): extended release dipyridamole 200mg/aspirin 25mg twice daily for 24 weeks
  Interventions: Drug: extended release dipyridamole 200mg/aspirin 25mg
- aspirin (Active Comparator): half a tablet of a 81mg aspirin twice daily for 24 weeks
  Interventions: Drug: 81mg aspirin

INTERVENTIONS:
Drug: extended release dipyridamole 200mg/aspirin 25mg — one tablet twice daily for 24 weeks
  Other Names: Aggrenox
  Arms: extended release dipyridamole/aspirin
Drug: 81mg aspirin — half a tablet twice daily for 24 weeks
  Other Names: ASA
  Arms: aspirin

SUMMARY:
Dipyridamole, a medication extensively used in combination with aspirin for stroke prevention, is a promising new treatment for lupus. Dipyridamole has been shown to inhibit certain lymphocyte populations that are over-reactive in lupus and to delay the emergence of lupus-related pathology in mice with lupus. The investigators are interested in investigating the efficacy of dipyridamole in preventing flares in patients with lupus and its impact on biomarkers of disease activity.

DETAILED DESCRIPTION:
T cells in systemic lupus erythematosus (SLE) express an abnormal phenotype characterized by increased effector functions and deficient regulatory responses. Dipyridamole, a phosphodiesterase inhibitor extensively used in combination with low dose aspirin in secondary stroke prevention, has been proposed as a specific T cell directed treatment for SLE. Dipyridamole inhibits the calcium/calcineurin/NF-AT pathway in SLE T cells in vitro and abrogates expression of cytokines and costimulatory molecules, eventually also affecting B cell responses. Dipyridamole delays the emergence of lupus related pathology in lupus prone mice, but has not yet been studied in humans with SLE. The investigators aim to investigate the efficacy of dipyridamole in the prevention of flares in SLE patients after withdrawal of background immunosuppressive medications. The investigators will additionally evaluate the safety and tolerability of dipyridamole and its impact on quality of life measures in this population. Furthermore, the effect of dipyridamole on T and B cell biomarkers will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SLE meeting the 1997 ACR Classification Criteria
* Evidence of positive ANA or anti-dsDNA within one year of screening
* SLEDAI ≥4 or ≥1 BILAG A or B at screening, despite standard of care

Exclusion Criteria:

* Leukopenia (WBC <2.000/mm3) or lymphopenia (lymphocytes < 300/mm3)
* AST or ALT >3 times above normal cut off values
* Acute lupus nephritis defined as class II, IV or V nephritis diagnosed within 6 months or prot/creat > 1.5 gm/gm due to active lupus or in process of receiving induction therapy for nephritis
* Active CNS lupus affecting mental status
* Pregnancy or breast feeding
* Current requirement for anticoagulation
* Contraindication to aspirin or dipyridamole, including history of recent or severe GI bleeding, hemoglobin <9 mg/dL, platelet count of <30,000 /mm3 or unstable platelet count
* Any other medical condition, whether or not related to lupus which, in the opinion of the investigator would render the patient inappropriate or too unstable to complete the study protocol
* Inability or unwillingness to understand and/or sign informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Thanou, MD, Principal Investigator — Oklahoma Medical Research Foundation
Locations (1):
- Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Those who wish access to this data may contact Joan Merrill at joan-merrill@omrf.org for further information
Supporting Information: Study Protocol
Time Frame: The data will be available on or before June 1 2021
Access Criteria: For de-identified data only: Please submit a two page request describing the research you wish to do and the investigators credentials and current employment. This will be reviewed by our cohort advisory board and IRB prior to release.

REFERENCES:
- [Background] Kyttaris VC, Zhang Z, Kampagianni O, Tsokos GC. Calcium signaling in systemic lupus erythematosus T cells: a treatment target. Arthritis Rheum. 2011 Jul;63(7):2058-66. doi: 10.1002/art.30353. PMID 21437870
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited from the Oklahoma Medical Research Foundation clinic after a full informed consent process.
Pre-assignment Details: There were no pre-assignment restrictions or procedures.
Period: Overall Study
Arm/Group | Extended Release Dipyridamole/Aspirin | Aspirin
Started | 13 | 5
Completed | 9 | 5
Not Completed | 4 | 0
Not completed — Adverse Event | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Release Dipyridamole/Aspirin | Aspirin | Total
Number analyzed (Participants) | 13 | 5 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.0) | 43.8 (12.9) | 44.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 9 | 4 | 13
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 5 | 18
Mean BILAG Score at Entry [Mean (Standard Deviation); unit: units on a scale] — The BILAG (Britiish Isles Lupus Assessment Group) index is commonly used in international SLE trials. It provides a discontinuous scale that assigns a score to each active organ system based on assessment of disease as mild (BILAG C) moderate (B) or severe (A). A global score is derived by assigning 12 points to each organ rated severe (A) 8 points for moderate (B) and 1 point for mild (C), adding these together. Thus, the total score is weighted by the severity of disease in each organ. Mean population scores at baseline are calculated for each group.
  units on a scale | 11.2 (4.4) | 10 (4.9) | 10.9 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: British Isles Lupus Assessment Group Index-based Combined Lupus Assessment (BICLA)
Description: This is a landmark measure of percentage of patients who meet response criteria. To meet the BICLA response measure a patient must, compared to baseline, have a decrease in all moderate or severe scores on the British Isles Lupus Assessment Group (BILAG) index by at least one severity grade (Severe disease (BILAG A score) must drop to at least moderate (B or better) and B must drop to at least mild (C or not present). Also, there must be no increase in any other BILAG organ scores, no increase in The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score, and no increase in the physician's global assessment (PGA) by more than 10% of the scale. Furthermore, there may no off protocol medication increases. Note on all scales mentioned a higher score signifies greater disease activity. Ranges on BILAG could be 0-108 but are rarely greater than 36. SLEDAI could range 0-105 but is rarely greater than 20. PGA 0-100 but rarely greater than 76.
Time Frame: 24 weeks
Population: Full Analysis Set was analyzed including all randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Release Dipyridamole/Aspirin | Aspirin
Number analyzed (Participants) | 13 | 5
Participants | 3 | 2

2. Secondary Outcome: Systemic Lupus Erythematosus Responder Index (SRI) 4
Description: This is a landmark analysis of percentage of patients who meet the following response criteria: Compared to baseline there must be a 4 point decrease in the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI), no increase in The British Isles Lupus Assessment Group (BILAG) Index score and no more of an increase in Physician's Global Assessment (PGA) than 10% of the scale. As assessed here, there must also be no off protocol increase in medications. All scales signify worsening disease when scores increase. Ranges on BILAG could be 0-108 but are rarely greater than 36. SLEDAI could range 0-105 but is rarely greater than 20. PGA 0-100 but rarely greater than 76.
Time Frame: 24 weeks
Population: Full analysis set of all randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Release Dipyridamole/Aspirin | Aspirin
Number analyzed (Participants) | 13 | 5
Participants | 3 | 2

3. Secondary Outcome: SRI Component Analyses: 4 Point Drop in SLEDAI
Description: This is a landmark analysis of percentage of patients who, compared to baseline, have a 4 point drop in the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI). A 4 point decrease signifies a clinically significant decrease in disease activity as reported in many studies and as commonly used as a clinical endpoint in trials. SLEDAI could range 0-105 but is rarely greater than 20.
Time Frame: 24 weeks
Population: Full Analysis Set of all randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Release Dipyridamole/Aspirin | Aspirin
Number analyzed (Participants) | 13 | 5
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Description: All adverse events were recorded in the medical record and compiled for analysis.
Arm/Group | Extended Release Dipyridamole/Aspirin | Aspirin
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/5
Other Adverse Events (participants affected / at risk) | 13/13 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release Dipyridamole/Aspirin (N=13) | Aspirin (N=5)
Hysterectomy (Reproductive system and breast disorders) | 0 (0) | 1 (1) — This patient had sudden schedule change for non-emergent hysterectomy during the trial. Intubation was complicated by pneumonia but that did not prolong hospitalization (reported as non serious AE).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release Dipyridamole/Aspirin (N=13) | Aspirin (N=5)
Gastroenteritis (Gastrointestinal disorders) | 8 (12) | 3 (3)
Upper Respiratory Infection (Infections and infestations) | 1 (2) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (4) — Described as several dizzy spells with two episodes of near fainting or fainting
Spider Bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Bladder Outlet Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chlamydia infectoin (Infections and infestations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
herpes zoster (Immune system disorders) | 1 (1) | 0 (0)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
neuralgia (Immune system disorders) | 1 (1) | 0 (0)
Sleep Disorder (Nervous system disorders) | 1 (2) | 0 (0) — At two different points in the study patient experienced insomnia and hypersomulence
urticaria (Immune system disorders) | 2 (2) | 0 (0)
sprained ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
weight loss (General disorders) | 1 (1) | 0 (0) — This was not associated with anorexia reported by patient but no cause found. It continued for a number of weeks but did was not reported to continue after that

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT01781611/Prot_SAP_000.pdf